CLINICAL TRIAL: NCT02039739
Title: Evaluation of Effectiveness and Safety of Orsiro™ in Routine Clinical Practice; A Multicenter, Prospective Observational Study
Brief Title: Orsiro™ Drug Eluting Stent in Routine Clinical Practice
Acronym: IRIS ORSIRO
Status: Completed | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); Biotronik Korea Co., Ltd (Industry)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2014-02
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Angioplasty, Transluminal, Percutaneous Coronary; Coronary Artery Disease
Keywords: Orsiro; Drug Eluting Stent; Routine Clinical Practice; Angioplasty, Transluminal, Percutaneous Coronary; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Orsiro™ Drug Eluting Stent
  Interventions: Device: Orsiro™ Drug Eluting Stent group

INTERVENTIONS:
Device: Orsiro™ Drug Eluting Stent group

SUMMARY:
The purpose of this study is to evaluate effectiveness and safety of Orsiro™ Drug Eluting Stent in Routine Clinical Practice

ELIGIBILITY:
Inclusion Criteria:

* Age 20 and more
* Intervention with Orsiro™ Drug Eluting Stent
* Agreed with written informed consent form

Exclusion Criteria:

* Intervention with Orsiro™ drug eluting coronary stent and other drug eluting stent at the same time
* Life expectancy of 1year and under
* Cardiac shock

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Orsiro™ Drug Eluting Stent
Sampling Method: Non-Probability Sample
Enrollment: 1007 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Composite event rate | 1YEAR

SECONDARY OUTCOMES:
ALL DEATH | 5YEAR
CARDIAC DEATH | 5YEAR
MYOCARDIAL INFARCTION | 5YEAR
Composite event of death or myocardial infarction | 5YEAR
Composite event of cardiac death or myocardial infarction | 5YEAR
Target Vessel revascularization | 5YEAR
Target Lesion revascularization | 5YEAR
Stent thrombosis | 5YEAR
  stent thrombosis as classified by an Academic Research Consortium
Stroke | 5YEAR
Procedural success | 3day
  defined as less than 30% residual stenosis at the completion of procedure without death or Q wave myocardial infarction or urgent revascularization
  participants will be followed for the duration of hospital stay, an expected average of 3days.

CONTACTS AND LOCATIONS:
Locations (18):
- South Korea (18):
  - Hallym University Sacred Heart Hospital, Anyang
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Dankook University Hospital, Cheonan
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Gangwon National Univ. Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Hospital, Incheon
  - Inje University Pusan Paik Hospital, Pusan
  - Pusan National University Yangsan Hospital, Pusan
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.